CLINICAL TRIAL: NCT00003900
Title: A Phase II Study of Irinotecan (CPT-11) and Docetaxel (Taxotere) in Patients With Recurrent Non-Small Cell Lung Cancer
Brief Title: Irinotecan With Docetaxel in Treating Patients With Recurrent or Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-982453; CDR0000067071 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-05-03 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irinotecan + docetaxel (Experimental): Patients receive irinotecan IV over 90 minutes immediately followed by docetaxel IV over 60 minutes on day 1. Treatment is repeated every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 5 years or until death.
  Interventions: Drug: docetaxel; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: docetaxel
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining irinotecan and docetaxel in treating patients who have recurrent or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate of previously treated patients with recurrent non-small cell lung cancer after treatment with irinotecan and docetaxel. II. Determine the toxicity of this regimen in these patients. III. Determine the overall survival in this patient population.

OUTLINE: Patients receive irinotecan IV over 90 minutes immediately followed by docetaxel IV over 60 minutes on day 1. Treatment is repeated every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 5 years or until death.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) Reconfirmation of NSCLC required only if complete response for greater than 1 year Measurable or evaluable disease Tumor shrinkage or stability for at least 4 weeks on initial chemotherapy CNS metastases allowed, if symptoms controlled for greater than 8 weeks after surgery or radiotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: 0-1 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal AST no greater than 2 times upper limit of normal (ULN) Renal: Creatinine no greater than 2.5 times ULN Cardiovascular: No New York Heart Association class III or IV heart disease Other: No active infection At least 5 years since any other prior malignancy except curatively treated basal or squamous cell skin cancer, carcinoma in situ, or other cancers No grade 2 or worse peripheral neuropathy No uncontrolled diabetes mellitus No other serious underlying disease Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No greater than 1 prior NSCLC chemotherapy regimen, excluding low dose cisplatin as a radiosensitizer No prior irinotecan or docetaxel At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy No prior radiotherapy to greater than 25% of bone marrow Surgery: See Disease Characteristics Other: No concurrent phenytoin, phenobarbital, or other anticonvulsants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1999-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 5 years

SECONDARY OUTCOMES:
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex A. Adjei, MD, PhD, Study Chair — Mayo Clinic
Locations (19):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Molina JR, Nikcevich D, Hillman S, Geyer S, Drevyanko T, Jett J, Verdirame J, Tazelaar H, Rowland K, Wos E, Kutteh L, Nair S, Fitch T, Flynn P, Stella P, Adjei AA. A Phase II NCCTG study of irinotecan and docetaxel in previously treated patients with non-small cell lung cancer. Cancer Invest. 2006 Jun-Jul;24(4):382-9. doi: 10.1080/07357900600705318. PMID 16777690